CLINICAL TRIAL: NCT05287269
Title: Importance of Ocular Coherence Tomography During Cataract Assessment
Brief Title: Ocular Coherence Tomography During Cataract Assessment
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2112020
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Cataract Senile; Macula Hole; Epiretinal Membrane; Age Related Macular Degeneration; Vitreomacular Traction
Keywords: cataract, macular pathology, ocular coherence tomography
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane; Macular Degeneration; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ocular Coherence Tomography — OCT images were recorded as a fast macular radial line scan with captured on either Heidelberg Spectralis (Heidelberg Engineering GmbH, Germany) or Topcon DRI Triton (Topcon Medical Systems inc. USA).
  Other Names: Swept Source ocular coherence tomography

SUMMARY:
Many patients will have underlying maculopathy present when undergoing cataract surgery, which are not visible on fundoscopy alone. Knowledge of this underlying pathology will allow an improved consenting process and discussion with the patient regarding the risks, visual prognosis and recovery following cataract surgery. Incidental findings in the fellow eye would also allow for improved diagnosis and management of these patients without adding significant additional time to specialist high volume cataract assessment clinics.

DETAILED DESCRIPTION:
The majority of anterior segment pathology may be diagnosed with simple slit lamp biomicroscopy, but posterior segment pathology may not be quite so obvious and can be missed on simple examination especially if a visually significant cataract is present impeding the view. There is also a degree of subjectivity from how much the cataract impairs the vision in comparison to the other elements of the optical pathway within the eye, and whilst there is no single way to evaluate this.

Optical coherence tomography (OCT) has been widely present in ophthalmology clinics since it's development 20 years ago although it is not commonly used in all units for the pre-operative assessment of patients referred for cataract surgery in high volume set ups such as the National Health Service (NHS) in the United Kingdom. There may still be reluctance to use OCT in a normal cataract assessment clinic as it may be perceived as an additional step that decreases time efficiency and increase financial investment in the services.

In this study we sought to investigate the prevalence of retinal pathology in the patient cohort, the comparison of subjective clinical slit lamp fundoscopy assessmenet with OCT findings and the co-incidental OCT findings in the fellow eye at the time of cataract assessment. OCT was chosen as the most efficient way to support clinicians in the assessment clinics, and to see if the addition of this step added value to the patient consultation and pre-operative assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for cataract surgery

Exclusion Criteria:

* Patients unable to attend the cataract assessment clinic
* Morbid patients who cannot be assessed on OCT or slit lamp

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This was a prospective cross-sectional study of 626 consecutive patients attending cataract assessment clinics at the Sussex Eye Hospital between 2/11/20 and 6/11/20. ]As part of work to decrease waiting times for patients in the wake of the first wave of COVID-19 pandemic and the shutdown of non-emergency services, a week of activity dedicated to cataract assessment was undertaken at Brighton & Sussex University Hospitals NHS trust between 2nd and 6th November 2020.
Sampling Method: Non-Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of occult macular pathologies in the eye referred for cataract surgery | During the cataract assessment clinic
  Comparison of slitlamp biomicroscopy fundus finding with ocular coherence tomography (OCT) scan of the macula

SECONDARY OUTCOMES:
Incidence of macular pathologies in the fellow eye | During the cataract assessment clinic
  Noting the incidence of macular pathologies noted on OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Brighton & Sussex University Hospitals NHS Trust, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided